CLINICAL TRIAL: NCT04353388
Title: Post Market Observational Study of ESId (MDW Hematology Parameter) for Early Sepsis Detection in the Emergency Department (US Hospitals) and Potential Reduction in Time to Antibiotics - Washington University
Brief Title: Sepsis Post Market Observational Study and Potential Reduction of Time to Antibiotics - Washington University
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C48392
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-07

CONDITIONS: Sepsis; Adult Disease; Severe Sepsis; Emergency Department
MeSH Terms: conditions — Sepsis; Disease; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CBC-Diff Monocyte Volume Width Distribution: Monocyte Volume Width Distribution (MDW) is part of the CBC with Differential
  Interventions: Diagnostic Test: CBC-DIFF Monocyte Volume Width Distribution (MDW)

INTERVENTIONS:
Diagnostic Test: CBC-DIFF Monocyte Volume Width Distribution (MDW) — MDW measurement will be used to detect sepsis. Results will not be used to manage patients.

SUMMARY:
The purpose of this study is to demonstrate that addition of the Monocyte Width Distribution (MDW) parameter to current standard of care improves a clinician's ability to recognize sepsis in the Emergency Department, resulting in earlier decision to administer antibiotics from time of ED presentation for sepsis patients (simulated primary endpoint), with concomitant reductions in length of stay and in-hospital mortality for those patients (secondary endpoints).

DETAILED DESCRIPTION:
The objective of this study is to develop a method for identifying sepsis patients from electronic health records (EHR) based on Sepsis-2 criteria. Sepsis patients will be identified using a Sepsis Definition which includes meeting SIRS score of ≥2 within 12 hours of ED presentation and any microbial testing ordered within 24 hours of ED presentation. The patient will be enrolled if it meets the Sepsis Definition and additional EMR data elements will be extracted to complete case report form. Furthermore, objectives include to confirm the clinical validity and performance of MDW in a control population of sepsis patients where MDW is measured but not reported to physicians. This study is an observational study which will simulate the decision impact of MDW on sepsis identification and patient management

ELIGIBILITY:
Inclusion Criteria:

* All race and ethnicities
* Presenting to the emergency department with suspicion of infection
* Whose assessment includes a CBC with differential
* Meets EMR Sepsis Definition

Exclusion Criteria:

* Pregnancy
* Prisoners
* Transfers from other ED
* Previously enrolled

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to the ED where a CBC-Diff has been ordered by standard of care
Sampling Method: Probability Sample
Enrollment: 1139 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Potential reduction of Time to Antibiotics | 12 hours after ED presentation
  Validate MDW's ability to reduce time to first antibiotics ordered by physician (decision to treat)-Simulated

SECONDARY OUTCOMES:
Performance | 12 hours after ED presentation
  Validate MDW's ability to identify incidence of patients diagnosed as Sepsis vs Non-Sepsis, including SIRS and milder forms of infection (non-SIRS) meeting Sepsis EMR definition of >=2 SIRS criteria within 12 hours of ED presentation and any microbial testing collected within 24 hours of triage in the ED

OTHER OUTCOMES:
Health & Economic Benefits for Time to Antibiotics - Simulated | 12 hours after ED presentation
  Determine MDW's ability to potentially reduced hospital stay using a simulated economic model
Health & Economic Benefits for Hospital Stay - Simulated | 12 hours after ED presentation
  Determine MDW's ability to potentially reduced Hospital stay, if applicable, using a simulated economic model
Health & Economic Benefits for Mortality - Simulated | 12 hours after ED presentation
  Determine MDW's ability to potentially reduced hospital morality, if applicable, using a simulated economic model
Health & Economic Benefits for ICU Stay - Simulated | 12 hours after ED presentation
  Determine MDW's ability to potentially reduced ICU stay, if applicable, using a simulated economic model

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Osborn, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States